CLINICAL TRIAL: NCT06569407
Title: The Effect of Online Training Program on Evidence-Based Practices on Nurses' Competencies for Evidence-Based Practices and Clinical Decision-Making Levels: A Randomized Controlled Trial
Brief Title: Education Program on Evidence-based Practices on Nurses' Competencies and Clinical Decision-Making Levels
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Seda Sariköse, Principal Investigator, Assistant professor, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024.227.IRB3.093
Record Dates: First submitted 2024-08-09; First posted 2024-08-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Evidence Based Practice
Keywords: Evidence Based Practice; Clinical Desicion Making; Educational Program; Online Training; Nurse; Randomized Controlled Trial; Educational Intervention

STUDY DESIGN:
Intervention Model Description: The study is planned as an open-label, randomized and controlled experimental research.
Who Masked: Participant
Masking Description: According to the randomization table, nurses who volunteered to participate in the study will be assigned to the experimental and control groups by the single-blinding method. Nurses will be assigned to the experimental and control groups. The randomization process was performed by a statistician other than the researcher and communicated to the researcher. A computer-aided simple randomization method was used to ensure a homogeneous distribution of the gro. For this purpose, 70 sets were created using the functions on the internet address "https://www.random.org/integer-sets".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group nurses working in the inpatient wards (Experimental): The nurses in the experimental group are expected to fill in the data collection tools (Introductory Information Form for Nurses, Evidence-Based Practice Competency Scale, Clinical Decision Making Scale in Nursing) before the education and then participate in the education about evidence-based practices on the online platform and fill in the data collection tools (Evidence-Based Practice Competency Scale, Clinical Decision Making Scale in Nursing and Education Evaluation Form) 20 days after the education.
  Interventions: Other: Online Educational Intervention
- Control group nurses working in the inpatient wards (Placebo Comparator): The nurses in the control group were expected to complete the data collection tools (Introductory Information Form for Nurses, Evidence-Based Practice Competency Scale, Clinical Decision Making Scale in Nursing) before the educational booklet was given and 20 days after the education.
  Interventions: Other: Educational Booklet

INTERVENTIONS:
Other: Online Educational Intervention — An educational program for EBP based on the online learning model was planned to be developed based on the literature and expert opinions. In the program, in line with the literature, the introduction to the EBP, the importance of EBP, EBP steps, clinical research question design in line with PICO, and introduction of EBP databases. It is planned to include topics such as literature search strategies, types of research, use of scientific research and evidence evaluation tools, introduction of clinical decision support systems, reflection of EBP on patient care and clinical decision-making processes, and it is planned to determine the final version of the education content with expert opinions. The program will include recorded videos, slides and documents for each module. The content of the program will be integrated into the Koç University Online Programs Platform by the experts working at Koç University Educational Technologies Unit.
  Other Names: Online education program and educational booklet for nurses on EBP
  Arms: Experimental group nurses working in the inpatient wards
Other: Educational Booklet — An educational booklet for EBP was planned to be developed based on the literature and expert opinions. The learning objectives and content of the educational booklet to be developed will be created by considering Bloom's taxonomy. In line with the literature, it is planned to include topics such as introduction to EBP, importance of EBP, evidence-based practice steps, clinical research question design in line with PICO, introduction of evidence-based databases, literature search strategies, research types, use of scientific research and evidence evaluation tools, introduction of clinical decision support systems, reflections of EBP on patient care and clinical decision-making processes, and finalization of the booklet topics with expert opinions.
  Other Names: An educational booklet for EBP
  Arms: Control group nurses working in the inpatient wards

SUMMARY:
This clinical trial aims to develop an online education program and an educational booklet for nurses on EBP and to compare the evidence-based competencies and clinical decision-making levels of nurses trained with these two methods.

Hypotheses of the Study Ho: There is no statistically significant difference between the nurses' competency levels who participated in the online education developed for evidence-based practices and those who were informed of the educational booklet.

H1. The nurses' competency levels who participated in the online education developed for evidence-based practices are statistically higher than those who were informed of the educational booklet.

Ho: There is no statistically significant difference between the clinical decision-making levels of nurses who participated in the online education developed for evidence-based practices and nurses who were informed with the educational booklet.

H1: The clinical decision-making levels of the nurses who participated in the online education developed for evidence-based practices are statistically higher than those informed with the educational booklet.

Participants will:

The nurses in the intervention group are expected to fill in the data collection tools (Introductory Information Form for Nurses, Evidence-Based Practice Competency Scale, Clinical Decision Making Scale in Nursing) before the education and then participate in the education about evidence-based practices on the online platform and fill in the data collection tools (Evidence-Based Practice Competency Scale, Clinical Decision Making Scale in Nursing and Education Evaluation Form) 20 days after the education.

The nurses in the control group were expected to complete the data collection tools (Introductory Information Form for Nurses, Evidence-Based Practice Competency Scale, Clinical Decision Making Scale in Nursing) before the education booklet was given and 20 days after the education.

DETAILED DESCRIPTION:
One of the specific highlights of this project is that nurses' competencies and clinical decision-making skills can be increased with an education program developed for EBP. In addition, the online education design of the education program in this project will facilitate the integration of education into orientation programs and in-service training for nurses working in institutions where healthcare services are provided. At the same time, the fact that the education program has an online design and consists of an online education that includes modules compatible with smartphones without time and space restrictions shows the original value of the study. Therefore, this study aims to develop an innovative and generalizable online education program for nurses at EBP, contribute to the literature, and indirectly reduce the cost of care and contribute to safe patient care.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who agree to participate in the study and work in inpatient wards will be included.

Exclusion Criteria:

* Nurses who do not agree to participate in the study and do not work in inpatient wards will not be included in the sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Clinical decision making levels of nurses | Measured before the education program and 20 days after the implementation of the education program.
  The Clinical Decision-Making in Nursing Scale (CDMNS): This scale was developed by Jenkins in 1983 in the USA to determine nursing students' clinical decision-making level based on their statements. Although the scale was developed by applying it to nursing students, it can also be applied to clinical nurses involved in patient care. Edeer and Sarıkaya, in 2015, conducted the Turkish validity and reliability study. The scale consists of 40 items and four sub-dimensions. The subscales of the scale are "exploring options and ideas", "investigating goals and values", "evaluating results", and "investigating knowledge and adopting new knowledge impartially". Each subscale consists of 10 items. 22 items on the scale are positively significant. The 18 negatively significant items are reverse coded. Each item on the scale is evaluated as 5: always, 1: never. The total Cronbach Alpha value of the scale was found to be 0.78.
Nurses' competencies for evidence-based practice | Measured before the education program and 20 days after the implementation of the education program.
  Evidence-based Practice Evaluation Competence Questionnaire (EBP-COQ). The scale was developed by Ruzafa-Martinez in 2013 to determine the competency levels of nurses and nursing students towards EBP-COQ, and its Turkish validity and reliability were conducted by Yildiz and Güngörmüş in 2016. The scale consists of three sub-dimensions and 25 items. The attitude sub-dimension of the scale consists of items 1-13, the skill sub-dimension consists of items 14-16, and the knowledge sub-dimension consists of items 20-25. The scale is a five-point Likert scale (1: Strongly disagree, 5: Strongly agree), and the minimum score is 25, and the maximum score is 125. Negative items are reverse-coded. A higher score on the scale indicates more self-perceived competence, knowledge, and skills towards EBP and a more positive attitude towards EBP. The total Cronbach Alpha value of the scale was found to be 0.82.

SECONDARY OUTCOMES:
Education Evaluation | Immediately after the intervention
  Education Evaluation Form: This form includes questions about the content of the education program, its implementation, end-of-education outcomes, and the opinions and suggestions of the participants to evaluate the education program to be developed. This form will be integrated into the Koç University Online Programs Platform, where the training will take place, and it can be accessed at the end of the program.

OTHER OUTCOMES:
Descriptive Informations | Measured before the education program.
  Descriptive Information Form for Nurses: This form was prepared based on the literature. It includes socio-demographic (age, gender, marital status) and professional information (duration of professional experience, unit of work, weekly working time, working style, training status for EBP, etc.) of nurses and consists of 16 questions in total.

CONTACTS AND LOCATIONS:
Overall Officials: SEDA SARIKOSE, RN, PhD, Study Director — Koc University School of Nursing
Locations (1):
- Koc University School of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data of the experimental study can be shared with the researcher's approval following ethical conditions. However, the individual data of the participants participating in the study cannot be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Through study completion, an average of 1 year
Access Criteria: The data of the experimental study can be shared with the researcher's approval following ethical conditions. However, the individual data of the participants participating in the study cannot be shared.

REFERENCES:
- [Background] Ruzafa-Martinez M, Lopez-Iborra L, Moreno-Casbas T, Madrigal-Torres M. Development and validation of the competence in evidence based practice questionnaire (EBP-COQ) among nursing students. BMC Med Educ. 2013 Feb 7;13:19. doi: 10.1186/1472-6920-13-19. PMID 23391040
- [Background] Yildiz E, Gungormus Z. The validity and reliability study of the Turkish version of the evidence based practice evaluation competence questionnaire. Nurse Educ Today. 2016 Oct;45:91-5. doi: 10.1016/j.nedt.2016.05.030. Epub 2016 Jun 7. PMID 27429412
- [Background] Jenkins, H. Perceptions of decision making among baccalaureate nursing students as measured by the clinical decision making in nursing scale. 1983. doctors of thesess, University of Maryland.
- [Background] Durmaz Edeer, A., Sarıkaya, A. Adaptation of Clinical Decision Making in Nursing Scale to Undergraduate Students of Nursing: The Study of Reliability and Validity. International Journal of Psychology and Educational Studies. 2015; 2(3): 1-9. https://doi.org/10.17220/ijpes.2015.03.001
- [Background] Wu Y, Brettle A, Zhou C, Ou J, Wang Y, Wang S. Do educational interventions aimed at nurses to support the implementation of evidence-based practice improve patient outcomes? A systematic review. Nurse Educ Today. 2018 Nov;70:109-114. doi: 10.1016/j.nedt.2018.08.026. Epub 2018 Aug 29. PMID 30179782